CLINICAL TRIAL: NCT06022250
Title: A Phase I Study to Evaluate The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of JS207 in Patients With Advanced Malignant Tumor
Brief Title: The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of JS207 in Patients With Advanced Malignant Tumor
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Collaborators: Sponsor GmbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JS207-001-I
Record Dates: First submitted 2023-08-23; First posted 2023-09-01 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Advanced Malignant Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JS207 (Experimental)
  Interventions: Drug: JS207

INTERVENTIONS:
Drug: JS207 — Patients will receive specific dose of JS207 via intravenous infusion.

SUMMARY:
This is a Phase I open-label, multicenter study to evaluate the safety, tolerability, pharmacokinetics (PK),Pharmacodynamic characteristics, immunogenicity and antitumor activity of JS207 in patients with advanced malignant tumor. The Recommended dose for phase II trial （RP2D） will be determined based on the safety, tolerability, pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced malignant tumor confirmed by histology or pathology, failed by standard treatment, no standard treatment or no standard treatment is applicable;
2. Eastern Cooperative Oncology Group (ECOG) 0 or 1;
3. Life expectancy ≥ 12 weeks;
4. At least one measurable lesion according to RECIST 1.1;
5. Adequate organ function;

Exclusion Criteria:

1. central nervous system metastasis；
2. There is a pleural, abdominal or pericardial effusion that is clinically symptomatic or requires repeated management (puncture or drainage, etc.)；
3. Images in screening showed that the tumor surrounded important blood vessels or had obvious necrosis and voids, and the investigators believed that it might cause bleeding risk；
4. The presence of severe, unhealed or open wounds, active ulcers, or untreated fractures；
5. A history of significant bleeding tendency or severe coagulopathy；
6. The presence of poorly controlled hypertension；

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2023-09-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity （DLT）、adverse event（AE） | 2 Years
  Incidence and severity of DLT, adverse events (AE), Abnormal changes in laboratory and other tests with clinical significance
Maximum tolerated dose (MTD),RP2D | 2 Years
  Maximum tolerated dose (MTD), Recommended dose for phase II trial

SECONDARY OUTCOMES:
Peak concentration（Cmax） | 2 years
  The highest plasma drug concentration that can be achieved after medication
Time to peak（Tmax） | 2 years
  After a single dose, the time of peak blood concentration
Elimination half life（t1/2） | 2 years
  The time it takes the blood to reduce the concentration of the drug to half
Progression free survival(PFS) | 2 years
  The time from first dose to Disease progression or death
Overall survival (OS) | 2 years
  The time from first dose to death from any cause
Immunogenicity | 2 years
  Incidence of Anti-Drug Antibody (ADA)
Objective response rate (ORR) based on Response Evaluation Criteria In Solid Tumors 1.1 (RECIST1.1) | 2 years
  Defined as the proportion of subjects who achieved partial response (PR) or complete response (CR)

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Cancer Hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No